CLINICAL TRIAL: NCT00288184
Title: Randomized Double-blinded, Placebo-controlled, Cross-over Trial of Allopurinol for the Treatment of Newly Diagnosed Essential Hypertension in Adolescents
Brief Title: Uric Acid in Essential Hypertension in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DK64587-DENA (completed); K23DK064587 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Experimental): Hypertensive children received both placebo and allopurinol in a cross over design.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Allopurinol adminsitered one 200mg capsule by mouth twice daily. Placebo capsule once daily during crossover
  Arms: Allopurinol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blinded, placebo controlled, crossover trial of allopurinol for the treatment of children with newly diagnosed essential hypertension.

DETAILED DESCRIPTION:
The study will be a double-blinded crossover trial. We will recruit 40 children between the ages of 12 and 18 years, from the pediatric renal and hypertension programs at Texas Children's Hospital. The study consists of four phases, a screening phase a treatment phase, an interim washout phase and a crossover phase.

The screening phase will last between 1 and 2 weeks. Patients will be provided with a digital blood pressure monitor with an appropriately sized cuff and be instructed to perform daily blood pressure measurements and keep a blood pressure log. This will detect severe hypertension that needs immediate attention and identify patients or families in which compliance problems likely to compromise data collection. Blood tests will be done to determine eligibility based on clinical laboratory parameters and 10ml of blood will be sent to the research laboratory for measurement of erythropoetin, ADMA, MCP-1 and possibly other modulators of vascular tone. Girls who are post-menarche will have a urine or serum pregnancy test. Prior to the initiation of any study procedures, informed consent and child assent (if appropriate) will be obtained from the participant and parents. Immediately prior to the initiation of the treatment or placebo phase 24-hour ambulatory blood pressure monitoring (ABPM #1) will be performed. Urinary nitrates and protein to creatinine ratio will be measured as surrogates for NOS activation and ongoing renal damage. At the end of the screening phase, eligible patients will be randomly assigned to either placebo or allopurinol for the active phase. Children will receive the other during the crossover phase. The purpose of this blinding is to remove either participant or investigator bias from the acquisition of the data.

Active Phase: The active phase will last six weeks and include a clinic visit on the first day of the phase, laboratory testing between day 4 and 7, and telephone contact halfway through the phase. At the clinic visit, patients will receive their study medication (allopurinol or placebo) in a bottle prepared by the investigational pharmacy. Subjects on allopurinol will receive 10 mg/kg divided bid (maximum of 400mg). Laboratory tests will be performed 4 to 7 days after starting the medication to screen for hepatic or bone marrow toxicity (AST, ALT, CBC) and serum uric acid. Evidence for toxicity will cause un-blinding and withdrawal from the study. The families will also be instructed to continue the daily blood pressure log started in the screening phase. Twenty-four-hour ABPM and end of phase laboratory tests including, hemoglobin, serum uric acid, erythropoetin, ADMA, MCP-1 and urinary nitrates will be performed at the conclusion of the active phase, prior to discontinuing the study medication for the washout phase.

Washout Phase: Upon completion of the ABPM at the end of the active phase, the study medication will be discontinued. The families will continue the home BP logs. The washout phase will end when either the child meets criteria for hypertension or two weeks have elapsed since completion of the previous phase.

Crossover Phase: The crossover phase will identical in procedures to the active phase except that the medication will be that which was not previously received.

Follow-up visit: Upon completion of both arms the subjects will have a final clinic visit. The laboratory tests will be repeated and if the third ABPM is not complete it will be initiated. Conventional antihypertensive therapy will be discussed and initiated if appropriate. Routine follow up will be established for management of the child's hypertension and other medical problems.

ELIGIBILITY:
Inclusion Criteria:

Males or females 12 to 18 years in age.

SBP or DBP greater than 95th percentile for age, gender and height

Diagnosis of primary hypertension after initial workup

No pharmacological therapy for hypertension in the past 12 months

Females must have a negative urine pregnancy test.

Parental or guardian consent and child subject assent

Exclusion Criteria:

Severe or poorly controlled hypertension as defined by SBP or DBP more than 20mmHg >95th percentile for age, gender and height or a history of hypertensive encephalopathy

Identified cause of secondary hypertension Renal transplant

Taking a calcineurin inhibitor, azathioprine or another nucleoside analogue medication (These medications have potentially serious drug interactions with Allopurinol.)

Currently receiving antihypertensive medication(s) or diuretic(s)

Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary or renal disease (These abnormalities would be expected to alter drug metabolism and increase the likelihood of medication side effects.):

Schwartz Formula GFR less than 60ml/min/1.73m2, AST/SGOT greater than 2 times the upper limit of normal* ALT/SGPT greater than 2 times the upper limit of normal* Total or direct bilirubin more than 2 times the upper limit of normal* Hemoglobin less than 9 gm/dl WBC less than 3.000/mm3 Platelet count less than 100,000/mm3 *age-adjusted normal range

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Ambulatory BP | three months
Casual Blood Pressure | three months

SECONDARY OUTCOMES:
plasma renin activity | three months
Systemic vascular resistance | three months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I. Feig, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Feig DI, Soletsky B, Johnson RJ. Effect of allopurinol on blood pressure of adolescents with newly diagnosed essential hypertension: a randomized trial. JAMA. 2008 Aug 27;300(8):924-32. doi: 10.1001/jama.300.8.924. PMID 18728266